CLINICAL TRIAL: NCT05460975
Title: Association of Sonographic Glandular Tissue Component With Breast Cancer Risk Among Women With Dense Breasts: A Prospective, Multinational Validation Study
Brief Title: Breast Cancer Risk From Sonographic Glandular Tissue Component (or International GTC Study)
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Principal Investigator, Seoul National University Hospital
Other Study IDs: Breast Cancer Risk
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Screening
Keywords: Breast cancer; Dense breast; Risk factors; Ultrasonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An international multicenter study to prospectively validate the association between sonographic GTC and subsequent breast cancer risk in women with dense breasts.

DETAILED DESCRIPTION:
Women with similarly dense breasts on mammography may have different subsequent risks of developing breast cancer due to varying degrees of lobular involution. Breast ultrasound (US) can assess the relative amount of glandular tissue component (GTC) to the fibrous stroma in dense breast parenchyma and can reflect the amount of terminal duct lobular units (TDLU) as seen in histology. In women with dense breasts on mammography, an association between high levels of sonographic GTC, defined as the percent of glandular tissue within fibroglandular tissue, and an increased risk of breast cancer was demonstrated in a retrospective single-center study of 8483 Korean women. The purpose of this international multicenter study is to prospectively validate whether sonographic GTC is associated with subsequent breast cancer risk and whether it can provide additional information beyond established risk factors. In this study, investigators will enroll 16164 women with dense breasts (BI-RADS density categories C and D on mammography) undergoing screening breast US using either an automated or handheld device. GTC will be assessed qualitatively as minimal, mild, moderate, or marked at the time of US interpretation and will be dichotomized into low (minimal or mild) versus high (moderate or marked). The primary outcome is a pathologic diagnosis of breast cancer, including invasive cancer and ductal carcinoma in situ (DCIS). Women are observed from 3 months after date of GTC assessment to breast cancer diagnosis or censoring as a result of death or end date of complete cancer capture. Covariate information will be obtained from self-report at the time of breast US examination and includes age, race/ethnicity, menopausal status, first-degree family history of breast cancer, breast density, history of benign breast biopsy, BMI, age at first live birth, and hormone replacement therapy (HRT) usage. The 5-year cumulative incidence of breast cancer by level of sonographic GTC will be compared based on marginal standardization with the predicted risk summed to a weighted risk according to the observed covariate distribution in the study population. The association of sonographic GTC with breast cancer risk will be estimated by using the Fine-Gray subdistribution hazards model to account for the competing risk of death. In addition, investigators will compare the discriminatory accuracy of the breast cancer surveillance consortium (BCSC) 5-year risk score and the BCSC model integrated with sonographic GTC.

ELIGIBILITY:
Inclusion Criteria

1. be ≥ 40 and <70 years old at time of US
2. No history of previous breast cancer including DCIS
3. have dense breasts (BI-RADS category C and D on mammography performed within 12 months of breast US) and negative/benign BI-RADS assessment categories on mammography (BI-RADS 1, 2)
4. undergoing screening breast US using either automated or handheld device

Exclusion Criteria

1. history of bilateral prophylactic mastectomy
2. history of bilateral foreign body injection
3. history of bilateral breast implants
4. history of bilateral breast reduction surgery or surgical excision
5. currently pregnant or breast feeding in the preceding 6 months
6. Known distant metastasis from other primary cancer

Ages: 40 Years to 69 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 16164 women
Sampling Method: Non-Probability Sample
Enrollment: 16164 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Incident breast cancer within 3 months to 7 years after the assessment of sonographic GTC | from 3 months to 7 years after the GTC assessment
  The 5-year cumulative incidence of breast cancer and hazard ratio by level of sonographic GTC using standardized risk

SECONDARY OUTCOMES:
Correlation of sonographic GTC with risk according to tumor type | from 3 months to 7 years after the GTC assessment
  Correlation of sonographic GTC with risk according to tumor type (DCIS vs. invasive cancer)
Correlation of sonographic GTC with breast cancer according to the breast US device | from 3 months to 7 years after the GTC assessment
  Correlation of sonographic GTC with breast cancer according to the breast US device (hand-held vs. automated)
The expected-to-observed (E/O) number of cancer diagnoses and concordance index (discriminatory accuracy) | from 3 months to 7 years after the GTC assessment
  The expected-to-observed (E/O) number of cancer diagnoses and concordance index (discriminatory accuracy) for the BCSC model (5-year risk score) and BCSC model integrated with sonographic GTC
Breast US diagnostic performance according to sonographic GTC | from the examination till 1 year after the GTC assessment
  Sensitivity, specificity, positive predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SH, Moon WK. Glandular Tissue Component on Breast Ultrasound in Dense Breasts: A New Imaging Biomarker for Breast Cancer Risk. Korean J Radiol. 2022 Jun;23(6):574-580. doi: 10.3348/kjr.2022.0099. No abstract available. PMID 35617993
- [Background] Lee SH, Ryu HS, Jang MJ, Yi A, Ha SM, Kim SY, Chang JM, Cho N, Moon WK. Glandular Tissue Component and Breast Cancer Risk in Mammographically Dense Breasts at Screening Breast US. Radiology. 2021 Oct;301(1):57-65. doi: 10.1148/radiol.2021210367. Epub 2021 Jul 20. PMID 34282967
- [Background] Acciavatti RJ, Lee SH, Reig B, Moy L, Conant EF, Kontos D, Moon WK. Beyond Breast Density: Risk Measures for Breast Cancer in Multiple Imaging Modalities. Radiology. 2023 Mar;306(3):e222575. doi: 10.1148/radiol.222575. Epub 2023 Feb 7. PMID 36749212